CLINICAL TRIAL: NCT02436876
Title: Phase 2a Randomized, Single-Blind, Placebo-Controlled, 12-week Escalating Dose Study to Assess the Safety, Tolerability and Clinical Activity of 3 Concentrations of Locally Applied MBN-101 to Infected Bone Sites
Brief Title: Study to Assess Safety and Clinical Activity of Local MBN-101 in Treatment of Infected Bone Sites
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Microbion Corporation (Industry)
Collaborators: University of Pennsylvania (Other); University of California, San Francisco (Other); Medpace, Inc. (Industry); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBN-101-201; W81XWH-12-2-0100 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2015-04-28; First posted 2015-05-07 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Bacterial Infection
Keywords: Osteosynthesis; Complications; Infection or Inflammation; Orthopedic; Device; Fracture; Osteomyelitis
MeSH Terms: conditions — Bacterial Infections; Infections; Inflammation; Fractures, Bone; Osteomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Cohort 1 (Experimental): Single, intra-wound local administration of MBN-101; dosage = 0.5 µg/cm2; randomized 3:1 with placebo
  Interventions: Drug: MBN-101; Other: Placebo
- Cohort 2 (Experimental): Single, intra-wound local administration of MBN-101; dosage = 1.5 µg/cm2; randomized 3:1 with placebo
  Interventions: Drug: MBN-101; Other: Placebo
- Cohort 3 (Experimental): Single, intra-wound local administration of MBN-101; dosage = 5.0 µg/cm2; randomized 3:1 with placebo
  Interventions: Drug: MBN-101; Other: Placebo

INTERVENTIONS:
Drug: MBN-101 — MBN-101 is a locally administered, anti-infective drug product
  Other Names: MBN-101 Drug Product
Other: Placebo — The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient
  Other Names: Diluent; Vehicle

SUMMARY:
This study evaluates the safety and clinical benefit of MBN-101 administered intraoperatively to osteosynthesis or osteomyelitis sites for patients diagnosed with an orthopedic infection, with or without orthopaedic hardware. Three quarters of the patients will receive MBN-101, while the other one quarter will receive placebo.

DETAILED DESCRIPTION:
Postoperative orthopaedic infections, particularly antibiotic-resistant infections, present a serious clinical challenge to surgeons and other treating physicians. These infections frequently involve implanted foreign materials (stabilizing orthopaedic hardware), making infection of these sites much more likely than if foreign materials were not involved. MBN-101 has broad spectrum antimicrobial activity against orthopaedic wound pathogens.

This is a randomized, single-blind, placebo-controlled, multi-center study to assess the safety and tolerability of escalating doses of MBN-101 to treat orthopaedic infections during revision surgery, (a) with or without orthopaedic hardware, and (b) with or without removal and replacement of orthopaedic hardware.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for this study, each of the following criteria must be satisfied with a "YES" answer (unless not applicable):

Patients who:

* have had operative fracture fixation of the upper extremity (AO/OTA class 15, 11-13, 21-23), lower extremity (AO/OTA class 31-34, 41 44, 81, 82) or pelvis (61, 62), or have undergone arthrodesis, and have subsequently been diagnosed with an apparent fracture site infection or are diagnosed with chronic or acute-on-chronic osteomyelitis of the long bone extremities (including residual amputated limbs)
* have at least one of the following:
* require surgical debridement of infected soft tissue and/or bone, with or without removal and/or placement/replacement of hardware
* male or female between the ages of 18 and 75 at the time the ICF is reviewed and signed
* patients receiving or anticipated to receive systemic antibiotic therapy as per institution's standard of care
* patients requiring postoperative hospitalization for at least 48 hours after revision surgery
* have read and signed the Informed Consent Form (ICF) after the nature of the study has been fully explained
* be willing and able to provide authorization for use and disclosure of personal health information in accordance with the Health Insurance Portability and Accountability Act (HIPAA)

Exclusion Criteria:

* To be eligible for this study, each of the following criteria must be satisfied with a "NO" answer (unless not applicable):

  * Patients who are no longer hardware dependent or are definitively treated for their infection by hardware removal without replacement
  * Patients with multiple, non-contiguous sites of infection
  * Pathologic fracture (not including osteoporosis)
  * Patient requires immunosuppressive therapy (Topical or inhaled corticosteroids are permitted)
  * Serum creatinine, ALT, AST or Alkaline Phosphatase >2.0 times the upper limit of the normal range of the local testing laboratory
  * Absolute neutrophil count <1000
  * Patients without definitive soft-tissue coverage over the surgical site at time of study product administration
  * Any condition that has required treatment with any other bismuth containing compound within the last 2 weeks (i.e., Kaopectate or Pepto Bismol)
  * Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months
  * Individuals undergoing surgical treatment for more than one infected site
  * Patients who are pregnant, lactating, or female patients who have a positive serum hCG (human Chorionic Gonadotropin) as determined by laboratory testing
  * Immunocompromised due to illness or organ transplant
  * History of chronic or recurrent infections (≥ 3 infections at the same site within 12 months)
  * History of any type of cancer (excluding non-melanomatous localized skin cancer or completely excised and cured carcinoma-in-situ of uterine cervix)
  * Poorly controlled diabetes mellitus
  * History of medical noncompliance
  * Other medical conditions which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results.
  * Current incarceration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Baker, MSc, DC, Study Chair — Microbion Corporation
Locations (6):
- United States (6):
  - Orthopedic Trauma Institute, University of California San Francisco, San Francisco, California
  - UCSF - Parnassus, San Francisco, California
  - LifeBridge Health, Inc., Baltimore, Maryland
  - OhioHealth Research Institute, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas - Health Science Center & Medical School at Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral. The study was sponsored by Microbion Corporation and conducted at 6 hospital clinical sites in the United States. The study was initiated on May 24, 2016, the Primary Completion Date was October 27, 2017, and the Study Completion Date was July 26, 2018.
Pre-assignment Details: A total of 20 patients were treated and completed the study.
Groups:
- MBN-101 0.5 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 0.5 µg/cm2; randomized 3:1 with placebo
  MBN-101: MBN-101 is a locally administered, anti-infective drug product
- MBN-101 1.5 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 1.5 µg/cm2; randomized 3:1 with placebo
  MBN-101: MBN-101 is a locally administered, anti-infective drug product
- MBN-101 5.0 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 5.0 µg/cm2; randomized 3:1 with placebo
  MBN-101: MBN-101 is a locally administered, anti-infective drug product
- Placebo: Placebo: The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient. Placebo subjects were randomized 1:3 with subjects treated with active.
Period: Overall Study
Arm/Group | MBN-101 0.5 µg/cm2 | MBN-101 1.5 µg/cm2 | MBN-101 5.0 µg/cm2 | Placebo
Started | 6 | 9 | 7 | 7
Treated | 6 | 6 | 6 | 7
Completed | 5 | 5 | 5 | 5
Not Completed | 1 | 4 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 2 | 1 | 0
Not completed — Inadequate amount of study drug available for randomization | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MBN-101 0.5 µg/cm2; MBN-101 1.5 µg/cm2; MBN-101 5.0 µg/cm2: Single, intra-wound local administration of MBN-101; randomized 3:1 with placebo
  MBN-101 is a locally administered, anti-infective drug product
- Total: Total of all reporting groups
Arm/Group | MBN-101 0.5 µg/cm2 | MBN-101 1.5 µg/cm2 | MBN-101 5.0 µg/cm2 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 6 | 6 | 21
  >=65 years | 2 | 1 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 2 | 8
  Male | 4 | 3 | 5 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 4
  White | 5 | 4 | 6 | 4 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This study evaluates the safety and tolerability of single escalating doses of locally administered MBN-101 or placebo, as adjunct to standard of care antimicrobial and surgical therapy.
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- MBN-101 0.5 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 0.5 µg/cm2; randomized 3:1 with placebo
- MBN-101 1.5 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 1.5 µg/cm2; randomized 3:1 with placebo
- MBN-101 5.0 µg/cm2: Single, intra-wound local administration of MBN-101; dosage = 5.0 µg/cm2; randomized 3:1 with placebo
- Placebo: The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient. Placebo was randomized 1:3 with active drug product treatment Cohorts 1-3
Arm/Group | MBN-101 0.5 µg/cm2 | MBN-101 1.5 µg/cm2 | MBN-101 5.0 µg/cm2 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7
participants
  Safety: TEAEs | 5 | 4 | 1 | 6
  Safety: Drug-related TEAEs | 1 | 1 | 1 | 1
  Safety: SAEs | 4 | 2 | 0 | 3

2. Secondary Outcome: Number of Treatment Failures
Description: Treatment failure is defined as clinical course requiring additional infection-related interventions including rehospitalization, additional surgery, or additional courses of systemic antibiotics.
Time Frame: 12 weeks
Measure: Number; unit: Treatment failure events
Groups:
- Placebo: Placebo: The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient. The placebo was randomized 1:3 with active drug product in Cohorts 1-3.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7
Treatment failure events | 1 | 2 | 1 | 3

3. Secondary Outcome: Treatment Failure in Subjects With Antibiotic-resistant Infections
Description: Treatment failure in subjects with baseline infections resistant to one or more antibiotics based on Central Laboratory Microbiological data
Time Frame: Up to 12weeks
Measure: Number; unit: Failures in antibiotic-resistant subject
Groups:
- Placebo: The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient. Placebo was randomized 1:3 with active drug product in Cohorts 1-3.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Placebo
Number analyzed (Participants) | 4 | 5 | 4 | 4
Failures in antibiotic-resistant subject | 1 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Placebo: Placebo: The placebo is comprised of the vehicle/excipients used to formulate MBN-101, but does not contain the active pharmaceutical ingredient. Placebo subjects were randomized 1:3 with subjects treated with active drug product in Cohorts 1-3.
Arm/Group | MBN-101 0.5 µg/cm2 | MBN-101 1.5 µg/cm2 | MBN-101 5.0 µg/cm2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/6 | 0/6 | 3/7
Other Adverse Events (participants affected / at risk) | 5/6 | 2/6 | 1/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBN-101 0.5 µg/cm2 (N=6) | MBN-101 1.5 µg/cm2 (N=6) | MBN-101 5.0 µg/cm2 (N=6) | Placebo (N=7)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This patient had significant underlying co-morbidities. A total of 10 non-drug-related SAEs were recorded. Not considered possibly or probably related to study drug (MBN-101 or placebo).
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Wound dehiscence (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Drug hypersensitivity (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — This was a drug hypersensitivity to a concommitant medication (Bactrim). Not considered possibly or probably related to study drug (MBN-101 or placebo).
Serious injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Road traffic accident causing multiple injuries. Not considered possibly or probably related to study drug (MBN-101 or placebo).
Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Deep vein thrombosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
C. difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Septic shock (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Linear Immunoglobulin A disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBN-101 0.5 µg/cm2 (N=6) | MBN-101 1.5 µg/cm2 (N=6) | MBN-101 5.0 µg/cm2 (N=6) | Placebo (N=7)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Increased measurement of systemic C-reactive protein (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Increased measurement of systemic red blood cell sedimentation rate (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) — Not considered possibly or probably related to study drug (MBN-101 or placebo).
Blood alkaline phosphatase increased (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) — Not considered possibly or probably related to study drug (MBN-101 or placebo) for one subject in the 0.5 µg/cm2 cohort, but possibly related to one subject in each of the 0.5 µg/cm2, 1.5 µg/cm2, 5.0 µg/cm2, and placebo cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT02436876/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT02436876/SAP_001.pdf